CLINICAL TRIAL: NCT04202562
Title: Efficacy and Safety of the ab Interno Trabeculectomy With Kahook Dual Blade Combined With Cataract Surgery Versus Cataract Surgery Alone: a Prospective, Single-center, Randomized Study
Brief Title: Efficacy and Safety of ab Interno Trabeculectomy With the Kahook Dual Blade
Acronym: KDB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Néstor Ventura Abreu, Medical Doctor, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16/560_P
Record Dates: First submitted 2019-12-15; First posted 2019-12-17 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension; Eye Diseases; Hypertension; Intraocular Pressure; Cataract
Keywords: Glaucoma; Ocular hypertension; Glaucoma, Open-Angle; Ab interno trabeculectomy; Phacoemulsification; Combined surgery; Minimally Invasive Glaucoma Surgery
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Eye Diseases; Hypertension; Cataract; Glaucoma | interventions — Cataract Extraction

STUDY DESIGN:
Intervention Model Description: One group received combined surgery, while the other cataract surgery alone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Combined surgery (Experimental): Participants intervened of combined ab interno trabeculectomy and cataract surgery at the same time
  Interventions: Procedure: Ab interno trabeculectomy; Procedure: Cataract
- Cataract surgery (Active Comparator): Participants intervened of cataract surgery alone
  Interventions: Procedure: Cataract

INTERVENTIONS:
Procedure: Ab interno trabeculectomy — Ab interno trabeculectomy performed after pupil contraction and 90 degrees ablation of the nasal trabecular meshwork
  Arms: Combined surgery
Procedure: Cataract — Cataract surgery with minimal clear cornea incision and phacoemulsification

SUMMARY:
The Kahook Dual Blade is a single-use device specially designed to create a clean cut in the trabecular meshwork. This ablation in the trabecular meshwork allows a better outflow of the aqueous humor, thus reducing the intraocular pressure (IOP), theoretically beyond the IOP reduction achieved by other minimally invasive glaucoma surgery (MIGS) devices.

Studies already published showed good results in terms of the reduction of the number of glaucoma medications and the reduction in the IOP, but not a single study has been performed prospectively comparing the efficacy of the technique, not even with the cataract surgery.

DETAILED DESCRIPTION:
This new device, the Kahook Dual Blade, has been specially designed to create a gentle cut compared to other cutting-devices that also remove the trabecular meshwork. Preclinical investigation showed no harm in the surrounding tissues. Only two prospective studies have been published, showing good results in terms of IOP reduction and a significant cut-off in the glaucoma medications. However, to better assess the real effect, a prospective comparison with cataract surgery or any other trabecular technique should be performed. We also aimed to determine the safety of the procedure.

Study design A prospective, randomized controlled, interventional study was conducted to determine the efficacy and safety of the Kahook Dual Blade. Patients with cataract and open-angle glaucoma or ocular hypertension (OHT) were included.

Subjects Patients were consecutively recruited from the Department of Glaucoma. Eligible patients were asked to participate if cataract surgery was indicated due to best-corrected visual acuity (BCVA) bellow 0.5 (in decimal scale), and moderate IOP reduction and a cut-off of the glaucoma medications was also aimed. Patients included in the study had been previously diagnosed with primary open-angle (POAG), pseudoexfoliative glaucoma (PSX) or OHT, and mild-to-moderate glaucoma according to the Hodapp-Parrish-Anderson classification, preoperative IOP ≤ 24 mmHg on at least one hypotensive medication, and coexistence of cataract without narrowing the angle (visible scleral spur at least in 2 quadrants). Both eyes from the same patient could be eligible if they both met the inclusion criteria.

Subjects who did not fulfill the inclusion criteria were excluded: patients with other glaucoma subtypes (elevated episcleral venous pressure, orbital occupancy, Sturge-Weber syndrome or any type of angle-closure glaucoma). Patients who underwent any intraocular surgery in the previous six months, including any laser or surgical intervention for glaucoma, or patients with any ophthalmic diseases that may interfere with tests were excluded. Severe or end-stage glaucoma or those with an indication of filtering or glaucoma drainage implant surgeries due to a high IOP with the maximum tolerated medication or glaucoma progression were also exclude.

All subjects were thoroughly examined before clinical intervention. This included a medical history review, slit-lamp examination, IOP determination with hand-held applanation tonometer, gonioscopy, dilated fundus examination, endothelial cell count (ECC) including cell and size automated detection with specular microscopy (EM-3000, Tomey Corporation, Nagoya, Japan), simulated keratometry (simK) determined by topography (Pentacam®, Oculus, Wetzlar, Germany), and standard automated perimetry (VF) (G1-Tendency Oriented Perimeter, Octopus® 1-2-3, Haag-Streit, USA).

Assignation and surgical technique For safety reasons, patients did not discontinue any topical hypotensive medications before surgery.

A randomized, controlled study was designed. Eyes were randomly assigned to each treatment group (www.random.org). If both eyes of the same patient were eligible to participate in the study, they could be allocated in different treatment groups due to randomization. All surgeries were performed by two experienced glaucoma surgeons. Standard cataract surgery with phacoemulsification using a 1.8 mm clear corneal incision (CCI) and intraocular lens (IOL) capsular bag placement was performed under topical anesthesia and 1% intracameral lidocaine. The surgeons were blinded to randomization until the end of the cataract surgery. At this point, if the patient was assigned to the treatment group the surgeon instilled acetylcholine 1% to reduce the pupillary size and facilitate visualization of the angle structures. To help maintain width, the anterior chamber was filled with a viscoelastic agent. Since the ab interno trabeculectomy is performed in the nasal quadrant, the surgeons then situated temporal, the patient's head was rotated 45 degrees in the opposite direction of the surgical site, and the microscope was tilted 30 to 45 degrees towards the surgeon. To guarantee better access to the nasal area of the angle, a 1.8 mm keratome was employed to widen the paracentesis. Further details of the surgical technique are described elsewhere.

Postoperative medications and follow-up Hypotensive medication was not administered intra- or post-operatively unless an IOP spike was detected. Postoperative topical treatment included a fixed combination of antibiotic plus steroid (tobramycin 0.3% and dexamethasone 0.1%) six times a day for seven days; this was tapered over the next four weeks.

Visits were undertaken at 1 day, 1 week, 1 month, 2 months, 3 months, 6 months, and 12 months. During follow-up, results of the slit-lamp examination, applanation tonometer IOP, and the number of medications were recorded at all visits. The VF and the ECC were also re-tested at 6 and 12 months. All the postoperative visits were conducted by the same examiner (NVA). Topical glaucoma medication was re-introduced if the target IOP according to the severity of the visual field was not achieved, o a higher than preoperative IOP was found.

Outcome measures - Data analysis Data obtained from each group were evaluated to determine the efficacy and safety of both interventions. The primary study outcomes were IOP and the number of glaucoma treatments. VF, ECC, BCVA and simK were secondary outcomes used to define the safety of both procedures. Success was defined as an IOP reduction of ≥ 20% from baseline; this cut-off was based on that reported in other glaucoma surgeries and is used for evaluation of this trabecular technique. The Saphiro-Wilk test was used to assess the sample distribution. Independent and dependent sample t-tests, when possible, were used to compare the results between groups and over time for each group. As both eyes of the same patient could be included in any of the treatment groups, generalized estimating equations (GEE) for repeated measures (IOP and number of medications) were also performed. A random-effect logistic regression was employed to analyse baseline characteristics associated with the success endpoint (IOP reduction of ≥20% from baseline). Statistical significance was set at a two-sided p-value ≤ 0.05. Statistical analyses were performed using Stata® version 14.1 (StataCorp, College Station, Texas, USA).

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 - 85 years
* Full comprehension and signing of the informed consent
* Preoperative intraocular pressure below 24 mmHg and at least one glaucoma medication
* Previous diagnose of open-angle glaucoma or ocular hypertension, including pseudoexfoliative glaucoma or pigment dispersion syndrome
* Mild to moderate glaucoma, according to the Hodapp-Parrish-Anderson classification

Exclusion Criteria:

* Not signing of the informed consent
* Not being able to attend to all the follow-up visits
* Young females during pregnancy or lactation
* Any other form of glaucoma not previously mentioned
* Glaucoma secondary to elevated episcleral venous pressure
* Preoperative best-corrected visual acuity lower than 0.1
* Clear lens extraction
* Severe or end-stage glaucoma
* Previous glaucoma surgery, cataract surgery or retinal surgery
* Patients taking anticoagulant medication that could not be discontinued during the perioperative period
* Oral anhydrase carbonic inhibitors
* Severe or uncontrolled systemic disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Evolution during follow up of the intraocular pressure | Up to 12 months
  in mmHg
Reduction in number of glaucoma medications | Up to 12 months
  Difference between number of glaucoma medications before and after the treatment

SECONDARY OUTCOMES:
Increase in visual acuity | Up to 12 months
  Best corrected visual acuity in decimal scale
Rate of reduction in endothelial cell count | Up to 12 months
  Number of cells, cells/mm^2
Increase of corneal astigmatism | Up to 12 months
  simulated keratometry, in diopters
Rate of visual field progression | Up to 12 months
  mean deviation, in decibels
Proportion of patients achieving the success endpoint | Up to 12 months
  Achieving a 20 percent reduction from basal intraocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: Julian Garcia Feijoo, Professor, Study Director — Hospital San Carlos
Locations (1):
- Hospital San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be shared if other investigators in their respective centers perform the clinical trial in a similar fashion. Personal information will not ever be shared, and medical records would be shared according to the current legislation of the European Union

REFERENCES:
- [Background] Greenwood MD, Seibold LK, Radcliffe NM, Dorairaj SK, Aref AA, Roman JJ, Lazcano-Gomez GS, Darlington JK, Abdullah S, Jasek MC, Bahjri KA, Berdahl JP. Goniotomy with a single-use dual blade: Short-term results. J Cataract Refract Surg. 2017 Sep;43(9):1197-1201. doi: 10.1016/j.jcrs.2017.06.046. PMID 28991617
- [Background] Dorairaj SK, Seibold LK, Radcliffe NM, Aref AA, Jimenez-Roman J, Lazcano-Gomez GS, Darlington JK, Mansouri K, Berdahl JP. 12-Month Outcomes of Goniotomy Performed Using the Kahook Dual Blade Combined with Cataract Surgery in Eyes with Medically Treated Glaucoma. Adv Ther. 2018 Sep;35(9):1460-1469. doi: 10.1007/s12325-018-0755-4. Epub 2018 Aug 4. PMID 30078175
- [Derived] Ventura-Abreu N, Garcia-Feijoo J, Pazos M, Biarnes M, Morales-Fernandez L, Martinez-de-la-Casa JM. Twelve-month results of ab interno trabeculectomy with Kahook Dual Blade: an interventional, randomized, controlled clinical study. Graefes Arch Clin Exp Ophthalmol. 2021 Sep;259(9):2771-2781. doi: 10.1007/s00417-021-05213-0. Epub 2021 Apr 27. PMID 33907888